CLINICAL TRIAL: NCT00403000
Title: Phase II Study of Dutasteride in Prostate Cancer Recurrent During Androgen Deprivation Therapy
Brief Title: Dutasteride in Treating Patients With Recurrent Prostate Cancer That Did Not Respond to Androgen-Deprivation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000514492; RPCI-I-34904
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dutasteride — Oral

SUMMARY:
RATIONALE: Dutasteride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well dutasteride works in treating patients with recurrent prostate cancer that did not respond to androgen-deprivation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the time to disease progression in patients with recurrent prostate cancer that progressed during androgen-deprivation therapy who are treated with dutasteride.
* Evaluate the toxicity of dutasteride in these patients.

Secondary

* Evaluate the serum prostate-specific antigen (PSA) level and objective radiographic response rate in patients treated with dutasteride.
* Determine the survival of patients treated with dutasteride.
* Determine the quality of life of patients treated with dutasteride.

OUTLINE: Patients receive oral dutasteride once daily until disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 3 months thereafter.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer

  * Asymptomatic progressive disease despite androgen-deprivation therapy

    * Progression must occur during androgen-deprivation therapy comprising orchiectomy or luteinizing hormone-releasing hormone (LHRH) analogue with or without antiandrogen AND after antiandrogen withdrawal

      * Concurrent LHRH monotherapy (i.e., LHRH analogs, such as leuprolide acetate or goserelin) required in patients who did not undergo prior bilateral orchiectomy to assure testicular androgen suppression
* Recurrent disease, as indicated by at least 1 of the following:

  * Prostate-specific antigen (PSA) at baseline ≥ 2.0 ng/mL
  * Biopsy-confirmed local recurrence
  * Increase in size of measurable lesions on radiographic study
  * New lesion on a nuclear bone scan
  * Two successive increases in serum PSA measured at least 1 week apart

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin ≤ 2.0 mg/dL
* SGOT ≤ 4 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 28 days since prior radiotherapy and recovered
* At least 28 days since prior flutamide OR at least 42 days since prior bicalutamide or nilutamide

  * Patients who have previously progressed despite antiandrogen withdrawal and who have started antiandrogens without reduction of serum PSA are eligible without requiring a 28- or 42-day washout interval after antiandrogen withdrawal
* No other prior systemic therapies, except androgen-deprivation therapy (i.e., orchiectomy or LHRH analogues only) or antiandrogens

  * Surgery, brachytherapy, external-beam radiotherapy, and cryotherapy are not considered systemic therapies
* No other concurrent anticancer therapy
* No concurrent use of any of the following:

  * Finasteride
  * Other investigational 5α-reductase inhibitors
  * Anabolic steroids
  * Alpha-receptor blockers (e.g., indoramin, tamsulosin hydrochloride, prazosin, terazosin, alfuzosin hydrochloride, and doxazosin)
  * Drugs with antiandrogenic properties (e.g., spironolactone, flutamide, bicalutamide, cimetidine, ketoconazole, metronidazole, and progestational agents)
  * Products containing selenium ≥ 75 mcg or vitamin E ≥ 100 IU
  * Saw palmetto
  * EG6761
* No concurrent radiotherapy, including palliative radiotherapy for pain control

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-12; Primary Completion 2007-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | Every 12 weeks
Toxicity | Daily while on Treatment

SECONDARY OUTCOMES:
Objective response (complete and partial) rate and serum prostate-specific antigen levels | Every 4 weeks
Survival | Every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James L. Mohler, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Shah SK, Trump DL, Sartor O, Tan W, Wilding GE, Mohler JL. Phase II study of Dutasteride for recurrent prostate cancer during androgen deprivation therapy. J Urol. 2009 Feb;181(2):621-6. doi: 10.1016/j.juro.2008.10.014. Epub 2008 Dec 16. PMID 19091347